CLINICAL TRIAL: NCT01614535
Title: Comparison of the Effect Site Concentration of Remifentanil for Preventing Cough During Emergence Between Male and Female Patients With Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4-2011-0356
Record Dates: First submitted 2012-06-03; First posted 2012-06-08 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Patients Undergoing Thyroidectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Female group (Experimental): Female gender patients undergoing thyroidectomy
  Interventions: Drug: up-and-down method to find out effective concentration of remifentanil for preventing cough during emergence
- Male group (Active Comparator): Male gender patients undergoing thyroidectomy
  Interventions: Drug: up-and-down method to find out effective concentration of remifentanil for preventing cough during emergence

INTERVENTIONS:
Drug: up-and-down method to find out effective concentration of remifentanil for preventing cough during emergence — Targeted effect-site TCI remifentanil for preventing cough effectively during emergence from general anesthesia. For effect-site TCI of remifentanil, a TCI pump was used and pump operation was based on Minto and colleagues' pharmacokinetic model. By Dixon's up-and-down method, the predetermined effect-site concentration(Ce) of remifentanil was determined according to the cough response of the previous patient. The initial target Ce of remifentanil for the first patient was 2.0 ng/ml. If the patients did not cough throughout the peri-extubation period, the predetermined Ce of remifentanil for the subsequent patient was decreased by 0.4 ng/ml. If the patient coughed anytime around extubation, the predetermined Ce for the subsequent patient was increased by 0.4 ng/ml. The stopping rule, as well as for the requirement of at least six turning points in the same direction of the sequential allocation response graph, required the recruitment of more than 20 patients.
  Other Names: remifentanil Ce, Ultiva Ce

SUMMARY:
The clinical studies demonstrate more powerful analgesic effect among female to both μ- and κ-opioid agonist (Fillingim et al. 2004). The antitussive effect of opioid is mediated predominantly by μ-, κ-opioid receptors (Kamei J. 1996). Therefore, the investigators hypothesized that there are sex differences in the antitussive responses to opioid.

It has been reported that target-controlled infusion (TCI) of remifentanil can reduce cough against endotracheal tube during emergence from general anesthesia. Some studies, reporting the EC50 and EC95 of remifentanil in effect-site TCI for preventing cough during emergence in different sex and surgeries (B. Lee et al. 2009, E.M.Choi et al. 2012), showed differences in EC50 and EC95.

The purpose of this study was to find out EC50 and EC95 of remifentanil in effect-site TCI for preventing cough during emergence in each sex and to evaluate whether there were sex differences in EC50 and EC95 of remifentanil in effect-site TCI or not.

ELIGIBILITY:
Inclusion Criteria:

* aged 20-46
* ASA classification I~II
* patients undergoing thyroidectomy

Exclusion Criteria:

* patient who has signs of a difficult airway
* patient who has smoking history
* patient who has upper respiratory infection or sore throat in the previous two weeks
* patient who has hypertension, DM
* female patients who were pregnant, breast-feeding or menopausal

Ages: 25 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
occurrence of cough | 20 minutes after sevoflurane off
  The cough was defined as a sudden contraction of the abdomen. The level of cough was assessed and recorded by the following cough grading system: Grade 0, no cough; Grade 1, single cough with mild severity; Grade 2, cough persistence less than 5 sec with moderate severity; Grade 3, severe, persistent cough for more than 5 sec.
  The patients will be followed from Sevolurane off to being transported to PACU.

CONTACTS AND LOCATIONS:
Overall Officials: Wyun Kon Park, MD, Principal Investigator — Yonsei University College of Medicine, Department of Anesthesiology and Pain Medicine
Locations (1):
- Department of Anesthesiology and Pain Medicine, Seoul, Seoul, South Korea